CLINICAL TRIAL: NCT02298946
Title: A Pilot Study of AMP-224, a PD-1 Inhibitor, in Combination With Stereotactic Body Radiation Therapy (SBRT) in Patients With Metastatic Colorectal Cancer
Brief Title: AMP-224, a PD-1 Inhibitor, With Stereotactic Body Radiation Therapy in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150021; 15-C-0021
Record Dates: First submitted 2014-11-21; First posted 2014-11-24 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma
Keywords: Anti-PD1 Therapy; Anti-Tumor Immunity; Liver Metastatic; B7-DC Fc Fusion Protein
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiosurgery; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DL1 - CTX, SBRTx1 day, & AMP-224 (Experimental): Dose Level 1 (DL1) Cyclophosphamide (CTX) 200mg/m(2) intravenous (IV) on day 0. Stereotactic body radiation therapy (SBRT) 8 (gray)Gy x 1 day on day 0, AMP-224 10mg/kg on day 1 then every (q)14 days for a total of 6 doses
  Interventions: Drug: AMP-224; Radiation: Stereotactic Body Radiation Therapy(SBRT); Drug: Cyclophosphamide
- DL2 - CTX, SBRTx3 days, and AMP-224 (Experimental): Dose Level 2 (DL2) CTX 200mg/m(2) IV on day 0, SBRT 8Gy x 3 day on days -2, -1, and 0. AMP-224 10mg/kg on day 1 then q14 days.
  Interventions: Drug: AMP-224; Radiation: Stereotactic Body Radiation Therapy(SBRT); Drug: Cyclophosphamide

INTERVENTIONS:
Drug: AMP-224 — 10mg/kg on day 1 then every 14 days for a total of 6 doses.
Radiation: Stereotactic Body Radiation Therapy(SBRT) — Dose Level 1: 8Gy x 1 day. Dose Level 2: 8Gy x 3 days
Drug: Cyclophosphamide — 200mg/m(2) IV on day 0.
  Other Names: CTX

SUMMARY:
Background:

- T-cells are white blood cells that can find and kill germs and tumors. Cancer can keep T-cells from working. Researchers think a new drug called AMP-224 might help the T-cells in people with cancer. They think the drug might work even better when combined with a certain type of radiation therapy.

Objective:

- To study the safety and effectiveness of AMP-224 together with 1 or 3 days of stereotactic body radiation therapy (SBRT) directed to the liver.

Eligibility:

- People age 18 and older with metastatic colorectal cancer. Their cancer must have spread to the liver and not be responding to treatment.

Design:

* Participants will be screened with a medical history, physical exam, and blood and urine tests. Their tumors will be measured with computerized tomography (CT) scans or magnetic resonance imaging (MRI) of the chest, stomach, and pelvis. They will have an electrocardiogram (ECG) heart test.
* Participants will have a small part of their tumor removed by needle (biopsy).
* Participants will have 8 study visits over about 10 weeks.
* At 1 visit, they will have another tumor biopsy.
* At 1 visit, they will get a chemotherapy drug through a vein (intravenous (IV)).
* At 6 visits, they will receive AMP-224 through an IV.
* At 1 or 3 visits, they will have SBRT. Computed tomography (CT) scans will map the position of their tumor. Radiation beams of different intensities at different angles will be directed to the tumor.
* At all visits, some screening procedures may be repeated.
* After treatment ends, participants will have 7 follow-up visits over about 5 months. Blood will be drawn. Some screening procedures may be repeated.

DETAILED DESCRIPTION:
Background:

* Colorectal cancer remains the second leading cause of cancer death in western countries with a median survival of approximately 24 months despite recent advances in systemic treatment.
* Several preclinical studies have documented an increase in peripheral antitumor immunity following radiation, a phenomenon known as the abscopal effect. Tumor PDL1 expression has also been shown to be induced by radiation, which can suppress the anti-tumor immune response. Inhibition of programmed cell death-1 (PD-1)/programmed death ligand-1(PDL-1) axis has been shown to improve anti-tumor immunity by blocking the tumor-mediated suppression of cytotoxic T cells.
* AMP-224, a B7-DC Fc fusion protein, binds to PD-1, an inhibitory receptor that is present on the cell surface of exhausted, activated, effector, and memory T cells. AMP- 224 has a unique mechanism of action in that it binds specifically to PD-1HI T cells (chronically stimulated / exhausted T cells) but not to PD-1LO cells which represent the normal activated T cells population
* The aim of the study is to evaluate whether the anti-tumor immunity of anti-PD1 therapy (with AMP-224) can be enhanced by radiation therapy.

Objectives:

- To assess safety, tolerability and feasibility of AMP-224 in combination with stereotactic body radiation therapy (SBRT) in patients with metastatic colorectal cancer.

Eligibility:

* Histologically confirmed metastatic colorectal cancer.
* Patient must have progressed on or been intolerant of prior oxaliplatin- and irinotecan containing regimen and have metastatic lesions that are not amenable to curative resection.
* Patient must have one focus of metastatic disease in the liver that is amenable to SBRT.
* Patient must have at least one measurable metastatic lesion by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria outside the radiation field.
* Patients must be willing to undergo mandatory pre and post treatment tumor biopsy.

Design:

* This is a pilot study whereby all patients will receive SBRT to one liver lesion and concomitant AMP-224. A single treatment of low dose/cyclophosphamide will be administered in conjunction with the SBRT therapy prior to the first AMP-224 treatment.
* Hypofractionated radiation will be administered to a metastatic disease site at a dose and schedule of 8Gy for 1 or 3 days in dose levels (DL)1 or 2 respectively. The day of first administration of AMP-224 will be designated as Day 1. In DL1 the SBRT will be administered on Day 0. In DL2 the SBRT will be administered from D-2 to D0. The study will begin with DL1 and escalate to DL2 once all subjects enrolled at DL1 have remained on study for 4 weeks, which is the DLT period.
* AMP-224 therapy will be given as an intravenous infusion beginning on Day 1 and then every 14 days for a total of 6 treatments only. Optional continuation of treatment q2- weekly until progressive disease (PD) will be considered in responding patients.
* Cyclophosphamide 200 mg/m(2) intravenous will be given on Day 0, prior to the first dose of AMP-224.
* Correlative studies: Peripheral blood will be collected (pre-dose) on days 1, 29, 57 and 93 for immune studies (including immunogenicity, circulating PD plasma samples, immune monitoring for phenotyping and peripheral blood mononuclear cells (PBMC) for T-cell activation). Tumor biopsies (formalin-fixed paraffin-embedded (FFPE) + Frozen) of an irradiated and non-irradiated liver lesion will be collected on day 1 and day 29, which will be analyzed by immunohistochemistry for tumor-infiltrating lymphocytes in addition to ribonucleic acid (RNA) analysis.
* Pharmacokinetic (PK) samples will be collected on Days 1, 15, 29, 43, 57, 71 in addition to up to 5 post treatment dates (if feasible).

ELIGIBILITY:
-Inclusion Criteria

1. Patients must have histopathological confirmation of Colorectal Carcinoma (CRC) by the Laboratory of Pathology of the National Cancer Institute (NCI) prior to entering this study.
2. Patients must have progressed on or been intolerant of prior oxaliplatin and irinotecan containing chemotherapeutic regimen and have disease that is not amenable to potentially curative resection. Patients who have a known KRAS wild type tumor must have progressed or been intolerant to cetuximab or panitumumab-based chemotherapy.
3. Patients must have one focus of metastatic disease in the liver that is amenable to stereotactic body radiation therapy (SBRT) in the opinion of radiation oncology.
4. All patients enrolled will be required to have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria outside the radiation field.
5. Study patients must have disease that is amenable to pre and post treatment biopsy and be willing to undergo this.
6. Age greater than or equal 18 years
7. Life expectancy of greater than 3 months
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
9. Patients must have acceptable organ and marrow function as defined below:

   * leukocytes less than or equal to 3,000/mcL
   * absolute neutrophil count less than or equal 1,500/mcL
   * platelets less than or equal 100,000/mcL
   * total bilirubin greater than or equal 1.5X institution upper limit of normal
   * Patients are eligible with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) measuring up to 5 x ULN given the presence of liver metastasis.
   * creatinine greater than 1.5X institution upper limit of normal

   Or

   -creatinine clearance less than or equal 45 mL/min/1.73 m(2), as calculated below, for patients with creatinine levels above institutional normal
10. Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1 or returned to baseline.
11. Patients must not have other invasive malignancies within the past 3 years (with the exception of non-melanoma skin cancers, localized prostate cancer, carcinoma in situ of the cervix and non-invasive bladder cancer that has had successful curative treatment).
12. Patient must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria

1. Prior immune checkpoint inhibition with anti-programmed cell death-1 (PD1)/programmed death ligand-1(PD-L1) or anti-cytotoxic T-lymphocyte antigen 4 (CTLA4) therapy or other specific T cell targeting agents.
2. Patients who have had chemotherapy (or so-called targeted systemic therapy), large field radiotherapy, or major surgery must wait 4 weeks after completing treatment prior to entering the study.
3. Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. Uncontrolled intercurrent illness including, but not limited to, hypertension (systolic blood pressure (BP) greater than 160, diastolic BP greater than 100), ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled diabetes or psychiatric illness/social situations that would limit compliance with study requirements.
5. Human immunodeficiency virus (HIV)-positive patients receiving anti-retroviral therapy are excluded from this study due to the possibility of pharmacokinetic interactions between antiretroviral medications and the investigational agent.
6. History of chronic autoimmune disease (e.g., systemic lupus erythematosus or Wegener's granulomatosis, Addison's disease, multiple sclerosis, Graves disease, Hashimoto's thyroiditis, hypophysitis, etc.) with symptomatic disease within the 3 years before randomization. Note: Active vitiligo or a history of vitiligo will not be a basis for exclusion. In addition, a past history of certain autoimmunity eg rheumatoid arthritis or thyroiditis may be allowed per principal investigator (PI) discretion provided it has been quiescent for a minimum of three years.
7. Active or history of inflammatory bowel disease (colitis, Crohn's), irritable bowel disease, celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea.
8. Dementia or significantly altered mental status that would prohibit the understanding or rendering of Information and Consent and compliance with the requirements of the protocol.
9. Currently receiving immunosuppressive doses of steroids or other immunosuppressive medications (inhaled and topical steroids are permitted)
10. History of sarcoidosis syndrome
11. History of hypersensitivity reaction to human or mouse antibody products.
12. Pregnancy and breast feeding are exclusion factors. The effects of AMP-224 on the developing human fetus are unknown. Enrolled patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, the duration of study participation and 3 months after the end of the treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
13. Patients with unhealed surgical wounds for more than 30 days.
14. Patients with known sensitivity or allergy to any components of AMP-224.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2016-07-13 (Actual); Study Completion 2017-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zitvogel L, Kepp O, Kroemer G. Immune parameters affecting the efficacy of chemotherapeutic regimens. Nat Rev Clin Oncol. 2011 Mar;8(3):151-60. doi: 10.1038/nrclinonc.2010.223. PMID 21364688
- [Background] Apetoh L, Ghiringhelli F, Tesniere A, Obeid M, Ortiz C, Criollo A, Mignot G, Maiuri MC, Ullrich E, Saulnier P, Yang H, Amigorena S, Ryffel B, Barrat FJ, Saftig P, Levi F, Lidereau R, Nogues C, Mira JP, Chompret A, Joulin V, Clavel-Chapelon F, Bourhis J, Andre F, Delaloge S, Tursz T, Kroemer G, Zitvogel L. Toll-like receptor 4-dependent contribution of the immune system to anticancer chemotherapy and radiotherapy. Nat Med. 2007 Sep;13(9):1050-9. doi: 10.1038/nm1622. Epub 2007 Aug 19. PMID 17704786
- [Background] Obeid M, Tesniere A, Ghiringhelli F, Fimia GM, Apetoh L, Perfettini JL, Castedo M, Mignot G, Panaretakis T, Casares N, Metivier D, Larochette N, van Endert P, Ciccosanti F, Piacentini M, Zitvogel L, Kroemer G. Calreticulin exposure dictates the immunogenicity of cancer cell death. Nat Med. 2007 Jan;13(1):54-61. doi: 10.1038/nm1523. Epub 2006 Dec 24. PMID 17187072
- [Derived] Floudas CS, Brar G, Mabry-Hrones D, Duffy AG, Wood B, Levy E, Krishnasamy V, Fioravanti S, Bonilla CM, Walker M, Morelli MP, Kleiner DE, Steinberg SM, Figg WD, Greten TF, Xie C. A Pilot Study of the PD-1 Targeting Agent AMP-224 Used With Low-Dose Cyclophosphamide and Stereotactic Body Radiation Therapy in Patients With Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2019 Dec;18(4):e349-e360. doi: 10.1016/j.clcc.2019.06.004. Epub 2019 Jul 2. PMID 31351862
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0021.html

RESULTS

PARTICIPANT FLOW:
Groups:
- DL1 - CTX, SBRTx1 Day, & AMP-224: Dose Level 1 (DL1) Cyclophosphamide (CTX) 200mg/m(2) intravenous (IV) on day 0, stereotactic body radiation therapy (SBRT) 8 (gray)Gy x 1 day on day 0, AMP-224 10mg/kg on day 1 then every (q)14 days
  AMP-224: 10mg/kg on day 1 then every 14 days for a total of 6 doses.
  Stereotactic Body Radiation Therapy(SBRT): Dose Level 1: 8Gy x 1 day Dose Level 2: 8Gy x 3 days
  Cyclophosphamide: 200mg/m(2) IV on day 0
- DL2 - CTX, SBRTx3 Days, and AMP-224: Dose Level 2 (DL2) CTX 200mg/m(2) IV on day 0, SBRT 8Gy x 3 day on days -2, -1, 0, AMP-224 10mg/kg on day 1 then q14 days
  AMP-224: 10mg/kg on day 1 then every 14 days for a total of 6 doses.
  Stereotactic Body Radiation Therapy(SBRT): Dose Level 1: 8Gy x 1 day Dose Level 2: 8Gy x 3 days
  Cyclophosphamide: 200mg/m(2) IV on day 0
Period: Overall Study
Arm/Group | DL1 - CTX, SBRTx1 Day, & AMP-224 | DL2 - CTX, SBRTx3 Days, and AMP-224
Started | 8 | 9
Completed | 4 | 8
Not Completed | 4 | 1
Not completed — Did not receive treatment | 2 | 0
Not completed — Unevaluable | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DL1 - CTX, SBRTx1 Day, & AMP-224 | DL2 - CTX, SBRTx3 Days, and AMP-224 | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (17.2) | 57.3 (14.5) | 58.8 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not meeting the definition for Hispanic or Latino | 7 | 9 | 16
  Mexican,Puerto Rican,Cuban,Central or So. Amer/Oth | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17
Count of Participants with Pre-Treatment Biopsies [Count of Participants; unit: Participants] | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 24 months and 8 days
Population: One patient (on dose level 1) after signing consent while waiting for radiation dosing, developed a spinal cord compression that needed emergent care at the local hospital. This patient was not treated. One patient (on dose level 1) after signing consent, developed a bowel obstruction prior to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 - CTX, SBRTx1 Day, & AMP-224 | DL2 - CTX, SBRTx3 Days, and AMP-224
Number analyzed (Participants) | 6 | 9
Participants | 6 | 9

2. Secondary Outcome: Duration of Response in Patients With Colorectal Cancer During and Following Treatment With AMP-224 in Combination With SBRT
Description: Duration of overall response is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is recorded first) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is complete disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: 12 months
Population: Zero participants were analyzed because no participants experienced a CR or PR.
Arm/Group | DL1 - CTX, SBRTx1 Day, & AMP-224 | DL2 - CTX, SBRTx3 Days, and AMP-224
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants in Which Specimens Were Collected for Pre and Post Pharmacokinetic (PK) AMP-224 Analyses
Description: This outcome measure only represents the number of participants with metastatic colorectal cancer who had specimens collected for pre and post pharmacokinetic (PK) AMP-224 analyses.
Time Frame: Baseline and post infusion AMP-224 (e.g. 15 minutes after infusion ended)
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 - CTX, SBRTx1 Day, & AMP-224 | DL2 - CTX, SBRTx3 Days, and AMP-224
Number analyzed (Participants) | 6 | 9
Participants
  Pre AMP-224 | 6 | 9
  Post AMP-224 | 6 | 9

4. Secondary Outcome: Overall Survival in Patients With Colorectal Cancer Following Treatment With AMP-224 in Combination With SBRT
Description: Overall survival is defined as the time from treatment start date until date of death or date last known alive.
Time Frame: Baseline to end of study, which is date of death. Average time participants were followed was 10.6 months.
Population: Patients were follow up post completion of the treatment medications for survival until date of their death. 2 patients were not evaluable since they did not receive treatment. 1 patient was lost to follow up after 3 cycles of treatment due to brain metastasis and treatment in another state.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DL1 - CTX, SBRTx1 Day, & AMP-224 | DL2 - CTX, SBRTx3 Days, and AMP-224
Number analyzed (Participants) | 6 | 9
months | 4.3 [1.2 to 8.9] | 9.0 [1.5 to 21.3]

5. Secondary Outcome: Count of Participants With Post-Treatment Biopsies
Description: Mandatory post treatment biopsies of the tumor were attempted on all patients.
Time Frame: Post treatment, day 29 +/- 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 - CTX, SBRTx1 Day, & AMP-224 | DL2 - CTX, SBRTx3 Days, and AMP-224
Number analyzed (Participants) | 8 | 9
Participants | 6 | 0

6. Secondary Outcome: Median Progression-free Survival in Patients With Colorectal Cancer
Description: Progression free survival is defined as the time interval from start of treatment to documented evidence of disease progression. Disease progression was evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: Baseline to disease progression, an average of 2.6 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DL1 - CTX, SBRTx1 Day, & AMP-224 | DL2 - CTX, SBRTx3 Days, and AMP-224
Number analyzed (Participants) | 6 | 9
months | 1.7 [0.9 to 3.3] | 2.7 [0.3 to 12.8]

7. Secondary Outcome: Objective Response Rate
Description: Objective response will be evaluated according to the revised Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and is defined as Complete Response + Partial Response. Briefly, complete response (CR) is defined as the disappearance of all target lesions, and Partial Response is defined as "at least" 30% decrease in the sum of the diameters of the target lesions from baseline measurement.
Time Frame: Restaging was done every 8 weeks for an average of 2.6 months.
Population: All patients had restaging evaluations completed as per protocol. Response criteria in solid tumors(RECIST) were completed on every trial participate. No partial or complete responses were found in any patients.
Measure: Number; unit: percentage of participants
Arm/Group | DL1 - CTX, SBRTx1 Day, & AMP-224 | DL2 - CTX, SBRTx3 Days, and AMP-224
Number analyzed (Participants) | 6 | 9
percentage of participants | 0 | 0

8. Secondary Outcome: Immunogenicity of AMP-224 as Measured by Human Anti-Murine Antibodies (HAMA) and Human Anti-Chimeric Antibodies (HACA) Concentrations
Description: Blood samples were collected to measure HAMA and HACA concentrations using the ELISA method in all patients.
Time Frame: Baseline, D1, D29, and D57 (pre-infusion), D79, D85 and 90 days post last dose (D169)
Population: Data was collected and not analyzed because the outside laboratory declined to run specimens with a negative clinical trial.
Arm/Group | DL1 - CTX, SBRTx1 Day, & AMP-224 | DL2 - CTX, SBRTx3 Days, and AMP-224
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Terminal Elimination Half-Life of AMP-224
Description: Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: 10 days
Population: as for outcome 8
Groups:
- All Participants: Dose Level 1 (DL1) Cyclophosphamide (CTX) 200mg/m(2) intravenous (IV) on day 0, stereotactic body radiation therapy (SBRT) 8 (gray)Gy x 1 day on day 0, AMP-224 10mg/kg on day 1 then every (q)14 days
  AMP-224: 10mg/kg on day 1 then every 14 days for a total of 6 doses.
  Stereotactic Body Radiation Therapy(SBRT): Dose Level 1: 8Gy x 1 day Dose Level 2: 8Gy x 3 days
  Cyclophosphamide: 200mg/m(2) IV on day 0 Dose Level 2 (DL2) CTX 200mg/m(2) IV on day 0, SBRT 8Gy x 3 day on days -2, -1, 0, AMP-224 10mg/kg on day 1 then q14 days
  AMP-224: 10mg/kg on day 1 then every 14 days for a total of 6 doses.
  Stereotactic Body Radiation Therapy(SBRT): Dose Level 1: 8Gy x 1 day Dose Level 2: 8Gy x 3 days
  Cyclophosphamide: 200mg/m(2) IV on day 0
Arm/Group | All Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Area of the Curve (AUC) of AMP-224
Description: The AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. The lower limit of quantification (LLOQ) is the smallest concentration of the drug that can be reliably measured.
Time Frame: Pre and post-infusion with all the AMP infusion and Day 1 at 8, 15, 29, 43, 57, and 71 hours.
Population: as for outcome 8
Arm/Group | DL1 - CTX, SBRTx1 Day, & AMP-224 | DL2 - CTX, SBRTx3 Days, and AMP-224
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of AMP-224
Description: Time maximum drug absorption is reached in the blood following administration of AMP-224.
Time Frame: 12.7 hours following intravenous (IV) infusion.
Population: as for outcome 8
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 24 months and 8 days.
Arm/Group | DL1 - CTX, SBRTx1 Day, & AMP-224 | DL2 - CTX, SBRTx3 Days, and AMP-224
All-Cause Mortality (participants affected / at risk) | 6/6 | 9/9
Serious Adverse Events (participants affected / at risk) | 4/6 | 2/9
Other Adverse Events (participants affected / at risk) | 6/6 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DL1 - CTX, SBRTx1 Day, & AMP-224 (N=6) | DL2 - CTX, SBRTx3 Days, and AMP-224 (N=9)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Death NOS (General disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) — malignant neoplasm
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DL1 - CTX, SBRTx1 Day, & AMP-224 (N=6) | DL2 - CTX, SBRTx3 Days, and AMP-224 (N=9)
Activated partial thromboplastin time prolonged (Investigations) | 5 (14) | 8 (19)
Alanine aminotransferase increased (Investigations) | 4 (6) | 3 (3)
Alkaline phosphatase increased (Investigations) | 4 (8) | 5 (8)
Anemia (Blood and lymphatic system disorders) | 5 (12) | 8 (16)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 4 (7)
Blood bilirubin increased (Investigations) | 3 (4) | 1 (1)
Blurred vision (Endocrine disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Edema limbs (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 4 (8) | 5 (6)
Fever (General disorders) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6) | 5 (7)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5) | 4 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 4 (8)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 3 (7) | 5 (12)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (8) | 8 (30)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 4 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (9) | 5 (10)
Pancreatic enzymes decreased (Investigations) | 1 (1) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) — urinary discomfort
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — outside CT scan, suggests pt might have pneumonia or increased lung lesion
Serum amylase increased (Investigations) | 1 (1) | 2 (4)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — diaphoresis
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT02298946/Prot_SAP_000.pdf
  • Informed Consent Form (2016-08-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT02298946/ICF_001.pdf